CLINICAL TRIAL: NCT04769323
Title: Use of Virtual Reality Devices for Vestibular Rehabilitation in Patients with Vestibular Hypofunction
Brief Title: Use of Virtual Reality Devices for Vestibular Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8
Record Dates: First submitted 2021-02-21; First posted 2021-02-24 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Virtual Reality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Group 1 use virtual reality.
  Interventions: Device: Virtual Reality
- Group 2 (Experimental): Group 2 do traditional home exercises.
  Interventions: Other: Traditional home exercises

INTERVENTIONS:
Device: Virtual Reality — Vestibular rehabilitation is an exercise-based program, designed by a specialty-trained vestibular physical therapist, to improve balance and reduce problems related to dizziness.
  Arms: Group 1
Other: Traditional home exercises — Vestibular rehabilitation is an exercise-based program, designed by a specialty-trained vestibular physical therapist, to improve balance and reduce problems related to dizziness.
  Arms: Group 2

SUMMARY:
The aim of this study is to investigate the superiority of virtual reality-supported vestibular rehabilitation exercises over conventional vestibular rehabilitation exercises in patients with complaints such as vertigo, loss of balance, falling, and gait imbalance.

ELIGIBILITY:
Inclusion Criteria:

* Complaining dizziness and/or instability for more than 3 months
* Patients aged 18 and over and under 65

Exclusion Criteria:

* Ear disease, head injury
* Ototoxic drug use
* Neurological and psychiatric illness that causes cooperation disorder
* Patients with orthopedic and systemic disorders that prevent exercising
* Patients with active malignancies
* Diseases that affect the use of glasses (epilepsy, vision loss, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-02-21 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Posturography | 1 year
  Posturography; It gives numerical data by comparing the data obtained from these three systems, whichever is caused by the patient's balance disorder, somatosensory system affected, visual system affected, or vestibular system affected.
Subjective Visual Vertical | 1 year
  Subjective visual vertical test, measures the functions of the utricular end organ.

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No